CLINICAL TRIAL: NCT03280615
Title: Effects of the Supplementation With Omega 3 Fatty Acids in Patients With Chronic Renal Disease
Brief Title: Omega 3 Fatty Acids in Patients With Chronic Renal Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Chile (Other)
Collaborators: Servicio de Salud Metropolitano Oriente (Unknown)
Responsible Party: Principal Investigator, Daniel Bunout, Full profesor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Omegarenal
Record Dates: First submitted 2017-08-08; First posted 2017-09-12 (Actual); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-07

CONDITIONS: Renal Insufficiency, Chronic
Keywords: Albuminuria; Carotid Intima-Media Thickness; Pulse Wave Velocity; Inflammation
MeSH Terms: conditions — Renal Insufficiency, Chronic; Albuminuria; Inflammation | interventions — Fatty Acids, Omega-3; Corn Oil

STUDY DESIGN:
Intervention Model Description: Participants will be randomly selected to receive 3.7 g of a supplement containing docosahexanoic and eicosapentanoic acids or a supplement containing corn oil. The supplements will be provided for 12 weeks
Who Masked: Participant, Care Provider, Investigator
Masking Description: Identical sachets containind the study supplement or corn oil will be number coded and provided to participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega 3 fatty acids (Experimental): Supplementation of 3.7 g of docosahexanoic and eicosapentanoic acids per day during 12 weeks
  Interventions: Dietary Supplement: Omega 3 fatty acids
- Corn oil (Placebo Comparator): Supplementation of 3.7 g of corn oil per day during 12 weeks
  Interventions: Dietary Supplement: Corn oil

INTERVENTIONS:
Dietary Supplement: Omega 3 fatty acids — Omega 3 fatty acids will be provided in a dose of 3.7 g/day, that should be enough to rise red blood cell levels of eicosapentanoic and docosahexanoic acids
  Arms: Omega 3 fatty acids
Dietary Supplement: Corn oil — Corn oil will be the placebo comparator for omega 3 fatty acids supplement
  Arms: Corn oil

SUMMARY:
To study the tolerance and efficacy of an omega 3 fatty acids supplement on renal and vascular function and inflammatory parameters in patients with chronic renal disease

DETAILED DESCRIPTION:
In a double blind trial in patients with chronic renal disease, the effects of a 3.7 g supplement of docosahexanoic and eicosapentanoic acids or a supplement of a similar dose of corn oil during 12 weeks, will be assessed on the following parameters:

1. Urine albumin excretion
2. Renal function measured with serum creatinine, cystatin C and beta-2 microglobulin
3. Carotid intima media thickness and pulse wave velocity
4. Inflammation status assessed measuring serum levels of C reactive protein and interleukin 6
5. Metabolic control of diabetes
6. Serum lipid levels

ELIGIBILITY:
Inclusion Criteria:

* Urinary albumin excretion over 30 mg/g creatinin
* Chronic renal failure stage 2 to 4
* Absence of serious conditions such as cáncer, decompensated heart failure, chronic infections and severe arterial lesions

Exclusion Criteria:

* Blood glucose levels over 180 mg/dl or glycosilated hemoglobin over 8%
* Presence of cognitive impairment that does not allow to sigin a written informed consent
* Alcohol or illicit drug abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Nutrition and Food Technology University of Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided
Sharing of information must be discussed with the sponsor

REFERENCES:
- [Background] Shapiro H, Theilla M, Attal-Singer J, Singer P. Effects of polyunsaturated fatty acid consumption in diabetic nephropathy. Nat Rev Nephrol. 2011 Feb;7(2):110-21. doi: 10.1038/nrneph.2010.156. Epub 2010 Dec 7. PMID 21135888
- [Background] Borg M, Svensson M, Povlsen JV, Schmidt EB, Aalkjaer C, Christensen JH, Ivarsen P. Long chain n-3 polyunsaturated fatty acids and vascular function in patients with chronic kidney disease and healthy subjects: a cross-sectional and comparative study. BMC Nephrol. 2016 Nov 21;17(1):184. doi: 10.1186/s12882-016-0393-5. PMID 27871238
- [Background] Xu T, Sun Y, Sun W, Yao L, Sun L, Liu L, Ma J, Wang L. Effect of omega-3 fatty acid supplementation on serum lipids and vascular inflammation in patients with end-stage renal disease: a meta-analysis. Sci Rep. 2016 Dec 23;6:39346. doi: 10.1038/srep39346. PMID 28008943
- [Background] Hoogeveen EK, Geleijnse JM, Kromhout D, Stijnen T, Gemen EF, Kusters R, Giltay EJ. Effect of omega-3 fatty acids on kidney function after myocardial infarction: the Alpha Omega Trial. Clin J Am Soc Nephrol. 2014 Oct 7;9(10):1676-83. doi: 10.2215/CJN.10441013. Epub 2014 Aug 7. PMID 25104273
- [Background] Malhotra R, Cavanaugh KL, Blot WJ, Ikizler TA, Lipworth L, Kabagambe EK. Dietary polyunsaturated fatty acids and incidence of end-stage renal disease in the Southern Community Cohort Study. BMC Nephrol. 2016 Oct 18;17(1):152. doi: 10.1186/s12882-016-0371-y. PMID 27756237

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omega 3 Fatty Acids | Corn Oil
Started | 50 | 50
Completed | 46 | 45
Not Completed | 4 | 5
Not completed — Lost to Follow-up | 1 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omega 3 Fatty Acids | Corn Oil | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67 [54 to 74] | 66 [56 to 74] | 66 [57 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 26 | 49
  Male | 27 | 24 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 50 | 50 | 100
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Chile | 50 | 50 | 100
Urine albumin excretion [Median (Inter-Quartile Range); unit: mg/g creatinine] | 363 [157 to 1030] | 541 [173 to 1125] | 455 [157 to 1079]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Urine Albumin Excretion Decrease of 20% or More
Description: Number of participants in whom urine albumin excretion in a spot urine sample at the end of follow up, expressed as mg/g creatinine, decreased by 20% or more
Time Frame: At baseline and 12 weeks of intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Omega 3 Fatty Acids | Corn Oil
Number analyzed (Participants) | 46 | 45
Participants | 19 | 13
Statistical Analysis 1: Comparison: Omega 3 Fatty Acids vs Corn Oil; A Fisher exact test was performed; Test type: Superiority; p = 0.257, Fisher Exact

2. Secondary Outcome: Change in C Reactive Protein Levels at 12 Weeks of Intervention
Description: Blood C reactive protein measured at baseline and the end of the intervention.
Time Frame: At baseline and 12 weeks of intervention
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Omega 3 Fatty Acids | Corn Oil
Number analyzed (Participants) | 46 | 45
mg/L
  baseline | 3.3 [1.5 to 5.3] | 1.7 [1.1 to 4.1]
  end of follow up | 2.1 [1.2 to 5.9] | 1.9 [1 to 5.2]
Statistical Analysis 1: Comparison: Omega 3 Fatty Acids vs Corn Oil; A mixed linear regression model for repeated measures was performed to test if the outcome behaved differently in both treatment groups; Test type: Superiority; p = 0.231, Fisher Exact

3. Secondary Outcome: Change in Pulse Wave Velocity at 12 Weeks of Intervention
Description: Measurement of pulse wave velocity using a oscillometric device measured at baseline and end of follow up and expressed ad m/s
Time Frame: At baseline and 12 weeks of intervention
Measure: Median (Inter-Quartile Range); unit: m/s
Arm/Group | Omega 3 Fatty Acids | Corn Oil
Number analyzed (Participants) | 46 | 45
m/s
  baseline | 9.8 [8.1 to 10.6] | 9.3 [8.5 to 10.7]
  end of follow up | 10.1 [8 to 10.9] | 9.7 [8.3 to 11.2]
Statistical Analysis 1: Comparison: Omega 3 Fatty Acids vs Corn Oil; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.043, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Three months of follow up
Arm/Group | Omega 3 Fatty Acids | Corn Oil
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 2/50 | 4/50
Other Adverse Events (participants affected / at risk) | 27/50 | 48/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omega 3 Fatty Acids (N=50) | Corn Oil (N=50)
Started dialysis (Renal and urinary disorders) | 2 (2) | 2 (2) — Started dialysis due to terminal renal failure
Hyperkalemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Cervical mass (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Cervical mass
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omega 3 Fatty Acids (N=50) | Corn Oil (N=50)
Nausea, vomiting or diarrhea (Gastrointestinal disorders) | 14 (14) | 12 (12)
Minor complaints (Product Issues) | 13 (13) | 36 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/15/NCT03280615/Prot_SAP_000.pdf